CLINICAL TRIAL: NCT03919006
Title: Levels of Netrin 1 and Its Receptor Unc5b in Gingival Crevicular Fluid, Saliva and Serum in Periodontal Disease and Health
Brief Title: Netrin 1 and Its Receptor Unc5b as Markers of Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Asst. Prof., Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017/87; 2018.06.05.1269 (Other Grant/Funding Number: Abant Izzet Baysal University Research Foundation)
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Periodontitis
Keywords: periodontal diseases; cytokines; gingival crevicular fluid; saliva; serum
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontitis (Active Comparator): GCF, saliva and serum samples were taken before and after treatment from periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment
- Gingivitis (Active Comparator): GCF, saliva and serum samples were taken before and after treatment from gingivitis patients.
  Intervention: Non- surgical periodontal treatment (Scaling and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment
- Periodontally healthy (Placebo Comparator): GCF, saliva and serum samples were taken at baseline from periodontally healthy individuals.
  Interventions: Other: Gingival crevicular fluid, saliva and serum collection

INTERVENTIONS:
Other: non surgical periodontal treatment — SRP under local anaesthesia, in a total of 2 clinical visits. Oral hygiene instructions including the modified Bass technique and an appropriate interdental cleaning device with dental floss and interdental brush.
  Arms: Gingivitis; Periodontitis
Other: Gingival crevicular fluid, saliva and serum collection — GCF with filter paper using the intracrevicular method, saliva and serum collection
  Arms: Periodontally healthy

SUMMARY:
This study aimed to investigate gingival crevicular fluid (GCF), saliva and serum Netrin 1 and Unc5b levels in periodontal health and disease. A total of 60 individuals, 20 patients with periodontitis, 20 with gingivitis and 20 periodontally healthy individuals were included. Whole-mouth and site-specific clinical periodontal parameters including probing depth, clinical attachment level, bleeding on probing, gingival index, plaque index and papillar bleeding index were recorded. GCF, salivary and serum Netrin 1 and Unc5b levels were measured by enzyme-linked immunosorbent assay. Statistical analysis was performed by using non-parametric tests.

DETAILED DESCRIPTION:
A total of 60 individuals, comprising 20 patients with Periodontitis (P Group), 20 patients with gingivitis (G Group), and 20 periodontally healthy controls (H Group) were involved in the study. The patients were diagnosed according to the new classification scheme. Stage and extent of periodontitis were also determined.

The clinical periodontal criteria for the diagnosis of the groups were as follows: the periodontitis group had interdental clinical attachment loss (CAL) ≥5 mm at site of greatest loss and periodontal probing depth (PD) ≥ 6 mm in one or more sites of the 2 non-adjacent teeth in at least two quadrants of the mouth. Accordingly, Stage III generalized periodontitis patients were included in the study. Patients were diagnosed as gingivitis with bleeding on probing ≥ 50 %, PD ≤3 mm, and no radiographic bone loss or CAL. Periodontally healthy individuals had no recorded history of periodontal problems, with PD ≤3 mm, no radiographic bone loss, good oral hygiene, no gingival inflammation.

Inclusion criteria were as follows: (1) aged >18 years, (2) having at least 16 natural teeth (excluding third molar),(3) nonsmokers with no history of smoking, (4) not having any diagnosed medical illness or drug intake that could affect the periodontal condition. The patients who had (1) taken antibiotics, nonsteroidal antiinflammatory or any other drugs within the past 3 months,(2) received nonsurgical or surgical periodontal treatment, (3) a restorative and endodontic therapy requirement, (4) a removable partial denture and/or having orthodontic therapy were excluded from the study. Current pregnancy or lactation and having serum C reactive protein (CRP) > 3mg/L were also the exclusion criteria.

All individuals were examined at baseline and four weeks after non-surgical periodontal treatment including, whole mouth probing depth (PD), CAL, presence of bleeding on probing (BOP), papillar bleeding index (PBI), gingival index (GI) and plaque index (PI) except the third molars. PD and CAL were measured at six sites per tooth using a manual periodontal probe.

The non-surgical periodontal treatment for periodontitis group included supra- and subgingival scaling, root planing and oral hygiene instructions. Subgingival scaling and root planing were performed under local anesthesia in two sessions within the 48-72 h. Gingivitis group had supra-and subgingival scaling, polishing and oral hygiene instructions. The treatment of gingivitis and periodontitis patients were performed by a periodontist (BM) using hand and ultrasonic instruments. All measurements were performed by the same calibrated examiner (SG).

Saliva sampling

Whole unstimulated saliva samples were collected. Each participant was asked first to rinse the mouth completely with tap water for 1 minutes, wait for 10 minutes, and then expectorate into sterile polypropylene tube for 5 minutes.

Gingival crevicular fluid (GCF) sampling

GCF samples were obtained from two nonadjacent interproximal sites in one single- rooted and one multi-rooted teeth by standardized filter paper strips. GCF was sampled from two sites with GI < 1, PD ≤ 3 mm and without BOP in the healthy group; two sites with GI ≥ 2, PD ≤ 3 mm and positive BOP (visible signs of inflammation) in the gingivitis group; and two deepest pocket (≥ 5 mm) with GI ≥ 2 and positive BOP in periodontitis group.

Serum sampling

Serum samples were taken following saliva and GCF sampling before the periodontal treatment. Six milliliters of venous blood were obtained by a standard venipuncture method and the serum was separated from blood by centrifugation at 1,500 g for 20 minutes.

Measurement of Netrin 1 and Unc5b levels in GCF, Saliva and Serum Samples

Netrin 1 and Unc5b levels in GCF, saliva and serum samples were measured by the enzyme-linked immunosorbent assay (ELISA) using commercial kits according to the manufacturer's guidelines.

Statistical Analysis

All data analyses were performed using a statistical software package. Comparisons of clinical and biochemical parameters between the study groups were performed using the Kruskal- Wallis with Mann Whitney U test with Bonferroni correction method. The intragroup comparisons (at baseline and first month) were performed using Wilcoxon test for paired samples. Associations among levels of the GCF, saliva and serum biomarkers and clinical parameters were also examined using the Spearman rank correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years,
* Having at least 16 natural teeth (excluding third molar),
* Nonsmokers with no history of smoking,
* Not having any diagnosed medical illness or drug intake that could affect the periodontal condition.

Exclusion Criteria:

* Patients who had taken antibiotics, nonsteroidal antiinflammatory or any other drugs within the past 3 months,
* Patients received nonsurgical or surgical periodontal treatment,
* Patients who have a restorative and endodontic therapy requirement,
* Having a removable partial denture and/or having orthodontic therapy,
* Current pregnancy or lactation and having serum CRP > 3mg/L .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (Netrin-1 and Unc5b) | Baseline and 4 weeks after treatment
  The changes in levels of Netrin-1 and Unc5b 4 weeks after periodontal treatment determined by ELISA.
  The changes in levels of Netrin-1 and Unc5b were analyzed to determine as a diagnostic biomarker of periodontal disease.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 4 weeks after treatment
  The changes in probing pocket depth was measured for determining severity of disease and clinical outcome
Clinical attachment loss | Baseline and 4 weeks after treatment
  The changes in probing pocket depth was measured for determining severity of disease
Gingival index | Baseline and 4 weeks after treatment
  Gingival index was recorded for classifying and evaluating sulcular gingival inflammation. Gingival index was also analyzed to detect the relationship between Netrin-1 and Unc5b.
Plaque index | Baseline and 4 weeks after treatment
  Plaque index was recorded for determining and classifying oral hygiene status
Bleeding on probing | Baseline and 4 weeks after treatment
  Bleeding on probing was recorded for classifying and evaluating gingival inflammation especially for apically sulcular inflammation. This was also analyzed to detect the relationship between Netrin-1 and Unc5b.
Papillar bleeding index | Baseline and 4 weeks after treatment
  Papillar bleeding index was recorded for classifying and evaluating the papillar gingival inflammation. This index was also analyzed to detect the relationship between Netrin-1 and Unc5b.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Asst. Prof., Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489